CLINICAL TRIAL: NCT01138475
Title: A Prospective, Randomized, Double-Blind, Double-Dummy,Placebo-Controlled, Parallel-Group, Pilot Trial Of Paricalcitol and Cholecalciferol(Vitamin D3) in the Treatment Of Secondary Hyperparathyroidism in Patients After ROUX-EN-Y Gastric Bypass Surgery
Brief Title: Trial Of Paricalcitol and Cholecalciferol(Vitamin D3) in the Treatment Of Secondary Hyperparathyroidism in Patients After ROUX-EN-Y Gastric Bypass Surgery
Acronym: ExtenD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kerstyn C. Zalesin, M.D. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Kerstyn C. Zalesin, M.D., Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-234
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2016-08

CONDITIONS: Gastric Bypass; Parathyroid Hormone
Keywords: PTH; Gastric bypass surgery; vitamin D; paricalcitol
MeSH Terms: interventions — paricalcitol; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paricalcitol (Active Comparator): This is a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules,cholecalciferol capsules, and matching placebo on PTH level at 6 weeks in patients with sHPT after RYGB. The pool of patients in the Beaumont Bariatric Surgery program will be sufficient to enroll approximately 75 subjects (25 per treatment group).
  Interventions: Drug: Paricalcitol
- cholecalciferol (Active Comparator): This is a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and matching placebo on PTH level at 6 weeks in patients with sHPT after RYGB. The pool of patients in the Beaumont Bariatric Surgery program will be sufficient to enroll approximately 75 subjects (25 per treatment group).
  Interventions: Drug: Cholecalciferol
- placebo (Placebo Comparator): This is a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and matching placebo on PTH level at 6 weeks in patients with sHPT after RYGB. The pool of patients in the Beaumont Bariatric Surgery program will be sufficient to enroll approximately 75 subjects (25 per treatment group).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — 1 microgram by mouth daily for 6 weeks
  Arms: Paricalcitol
Drug: Cholecalciferol — 5000 IU (international units) by mouth daily for 6 weeks
  Arms: cholecalciferol
Drug: Placebo — Inactive substance, one capsule daily for 6 weeks
  Arms: placebo

SUMMARY:
Evaluate the efficacy of paricalcitol, cholecalciferol, and placebo in the reduction of parathyroid hormone in patients after Roux-en-Y gastric bypass surgery (RYGB). Assess changes, if any, in measures of self-assessed well-being attributable to paricalcitol after RYGB. Evaluate the rates of hypercalcemia, kidney stones, gastrointestinal side effects, and other organ system adverse effects of paricalcitol, cholecalciferol, and placebo in patients after RYGB

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.

  2. Must be post bariatric (> 6 weeks and ≤ 5 years) Rou-en-Y gastric bypass surgical patient.

  3. Male or female subjects > 18 years. 4. For entry into the Treatment Period the subject must satisfy the following criteria based on the existing laboratory values previously drawn on clinical grounds:
  * Serum calcium level 8.0-10.5 mg/dL
  * Phosphorous level < 5.2 mg/dL (1.68 mmol/L)
  * Serum albumin > 3.0 g/dL (30 g/L). 5. For entry into the Treatment Period the subject must satisfy the following criteria based on screening laboratories (Beaumont Reference Laboratories, screening laboratory values are not blinded):
  * iPTH > 69 pg/ml
  * Negative serum pregnancy test for female subjects of childbearing potential. 6. In the opinion of the investigator, the subject must be receiving optimal medical management of other co morbidities including but not limited to HTN, DM, CVD, liver disease, and lung disease.

    7. If female, subject is not breast feeding or is not pregnant (verified by negative pregnancy test prior to the Treatment Period); or is not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy); or is of childbearing potential and practicing one of the following methods of birth control:
  * Double-barrier method (any two of the following: condoms, contraceptive sponge, diaphragm, vaginal ring with spermicidal jellies or creams, or intrauterine device [IUD])
  * Hormonal contraceptives (oral, parenteral, or transdermal) for at least three months prior to and during study drug administration
  * Maintains a monogamous relationship with a vasectomized partner
  * Total abstinence from sexual intercourse during the study (minimum one complete menstrual cycle prior to study start)

Exclusion Criteria:

* . Subject has previously been on active vitamin D therapy (calcitriol, paricalcitol, doxercalciferol, alfacalcidol) within the 30-day washout period prior to the Treatment Period at doses greater than 1200 IU of vitamin D3 or equivalent.

  2. Subject has a history of an allergic reaction or significant sensitivity to paricalcitol or to drugs similar to the study drug (i.e., vitamin D or vitamin D related compounds).

  3. Pregnant (confirmed by screening pregnancy test) or lactating females. 4. Subject is expected to initiate renal replacement therapy within one year. 5. Known history of hypercalcemia (>10.5 mg/dl), hyperphosphatemia (>6 mg/dl) primary hyperparathyroidism, or history of end-stage renal disease requiring renal replacement therapy.

  6. Full remission from a malignancy for less than one year (except completely excised non-Melanoma skin cancer e.g., basal or squamous carcinoma) or any history of bone metastasis.

  7. Subject has co-morbid conditions (e.g., advanced malignancy, advanced liver disease) with a life expectancy less than 1 year.

  8. Subject has received any investigational drug within 30 days prior to study drug administration or is currently enrolled in another clinical trial.

  9. Subject has a history of active kidney stones within the 2 years prior to the Screening Period.

  10. Subject has poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg at the Screening Visit (confirmed by repeat).

  11. Subject has history of renal artery stenosis, primary aldosteronism or pheochromocytoma, 12. Subject is taking calcitonin, bisphosphonates, cinacalcet, glucocorticoids (except topical or inhaled glucocorticoids), or other drugs that may affect calcium or bone metabolism, other than aluminum, calcium and non-calcium containing phosphate binders or female subjects on stable (same dose and product for three months) estrogen and/or progestin therapy.

  13. Subject is currently receiving immunosuppressant therapy and/or high doses (non-maintenance therapy) of glucocorticoids (> 5 mg/day of prednisone or equivalent).

  14. Subject has had acute renal failure within 12 weeks of the Screening Phase defined by an acute rise in serum Cr (of at least 0.5 mg/dL or 44 micromoles/L) to more than 4 g/dL (350 micromoles/L).

  15. Subject is known to be HIV positive. 16. Use of known inhibitors (i.e., ketoconazole) or inducers (i.e., carbamazepine) of cytochrome P450 3 A (CYP3 A) within two weeks prior to study drug administration.

  17. For any reason, subject is considered by the Investigator to be an unsuitable candidate to receive paricalcitol capsules or is put at risk by study procedures.

  18. Subject has a history of drug or alcohol abuse within six months prior to screening.

  19. Subject has had a liver or kidney transplant. 20. Stage V CKD subjects on renal replacement therapy are explicitly excluded. 21. Subject has had a CVA within the last 3 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerstyn Zalesin, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Health Center, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects have been recruited from our patients who underwent gastric bypass surgery. They needed to be able to give informed consent, age > 18 years, within 12 months of RYGB being performed, post-operative iPTH >69 pg/ml negative serum pregnancy test, serum calcium 8.0-10.5 mg/dl, phosphorus level <5.2 mg/dl, and serum albumin >3.0 g/dl.
Groups:
- Placebo-controlled: The placebo group received a placebo capsule, 1 daily each day of the week. This was a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and placebo on serum PTH levels after a 6-week trial in patients with secondary hyperparathyroidism after GB surgery. We enrolled 49 subjects (16, 17, and 16 in the paricalcitriol, cholecalciferol, and placebo groups, respectively).
  Consenting adult participants were randomized in a 1:1:1 ratio to each treatment group and received paricalcitol capsules, cholecalciferol capsules, or placebo. Per inclusion criteria, all had previously undergone GB for the treatment of morbid obesity, were between 6 weeks and 5 years post-surgery with secondary hyperparathyroidism, defined as a serum PTH level greater than 69 pg/mL.
- Paricalcitrol: Paricalcitriol arm received1 mcg daily each day of the week. This study was randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and placebo on serum PTH levels after a 6-week trial in patients with secondary hyperparathyroidism after GB surgery. We enrolled 49 subjects (16, 17, and 16 in the paricalcitriol, cholecalciferol, and placebo groups, respectively).
- Cholecalciferol: The cholecalciferol arm was treated with 5000 IU of cholecalciferol total of 35,000 IUper week.
  This study was randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and placebo on serum PTH levels after a 6-week trial in patients with secondary hyperparathyroidism after GB surgery. We enrolled 49 subjects (16, 17, and 16 in the paricalcitriol, cholecalciferol, and placebo groups, respectively).
Period: Overall Study
Arm/Group | Placebo-controlled | Paricalcitrol | Cholecalciferol
Started | 16 | 16 | 17
Completed | 16 | 16 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Cholecalciferol | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 16 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 16 | 49
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9) | 55 (10) | 51 (11) | 53.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 15 | 41
  Male | 1 | 6 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 17 | 49
PTH [Mean (Standard Deviation); unit: ng/mL] — Population: failure to capture
  ng/mL
    number analyzed (Participants) | 15 | 16 | 14 | 45
    (all) | 96 (27) | 90 (15) | 101 (25) | 96 (24)
alkaline phosphatase [Mean (Standard Deviation); unit: u/L] | 87 (19) | 97 (29) | 101 (32) | 95 (27)
serum calcium [Mean (Standard Deviation); unit: mg/dL] | 9.4 (0.3) | 9.3 (0.3) | 9.4 (0.4) | 9.3 (0.3)
25 OH vitamin D [Mean (Standard Deviation); unit: ng/dL] | 30 (16) | 32 (13) | 30 (7) | 30 (12)
serum phosphorous [Mean (Standard Deviation); unit: mg/dL] — Population: failure to capture
  mg/dL
    number analyzed (Participants) | 15 | 16 | 15 | 46
    (all) | 3.9 (0.6) | 3.7 (0.5) | 3.7 (0.5) | 3.7 (0.5)
24 hour urine calcium [Mean (Standard Deviation); unit: mmol] — Population: failure to capture
  mmol
    number analyzed (Participants) | 15 | 15 | 16 | 46
    (all) | 89 (81) | 106 (139) | 131 (91) | 109 (105)
osteocalcin [Mean (Standard Deviation); unit: ng/mL] — Population: failure to capture
  ng/mL
    number analyzed (Participants) | 14 | 15 | 16 | 45
    (all) | 39 (19) | 36 (17) | 40 (20) | 39 (19)
Urine N-telopeptide cross linked [Mean (Standard Deviation); unit: nmol] — Population: failure to capture
  nmol
    number analyzed (Participants) | 15 | 14 | 16 | 45
    (all) | 64 (26) | 73 (30) | 82 (55) | 73 (40)
bone specific alkaline phosphatase [Mean (Standard Deviation); unit: U/L] — Population: failure to capture
  U/L
    number analyzed (Participants) | 15 | 15 | 16 | 46
    (all) | 15 (5) | 19 (8.1) | 19 (10) | 18 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure With iPTH
Description: Change in iPTH was compared in each arm from baseline to final measure at 6 weeks the differences were compared in the 3 arms of the study
Time Frame: 6 weeks
Population: missing data in paricalcitol and placebo group
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Paricalcitol: This is a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules,cholecalciferol capsules, and matching placebo on PTH level at 6 weeks in patients with sHPT after RYGB. The pool of patients in the Beaumont Bariatric Surgery program
  Paricalcitol: 1 microgram by mouth daily for 6 weeks
- Cholecalciferol: This is a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and matching placebo on PTH level at 6 weeks in patients with sHPT after RYGB. The pool of patients in the Beaumont Bariatric Surgery program
  Cholecalciferol: 5000 IU (international units) by mouth daily for 6 weeks
- Placebo: This is a randomized, double-blind, double-dummy, placebo-controlled trial investigating the effects of paricalcitol capsules, cholecalciferol capsules, and matching placebo on PTH level at 6 weeks in patients with sHPT after RYGB. The pool of patients in the Beaumont Bariatric Surgery program
  Placebo: Inactive substance, one capsule daily for 6 weeks
Arm/Group | Paricalcitol | Cholecalciferol | Placebo
Number analyzed (Participants) | 15 | 17 | 15
pg/mL | 72 (31) | 87 (43) | 82 (30)

2. Secondary Outcome: Alkaline Phosphatase
Description: This secondary outcome measure is change in alkaline phosphatase from baseline to final measure at 6 weeks differences were compared between the 3 arms of the study
Time Frame: 6 weeks
Population: missing 1 participant data in the paricalcitol group
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Paricalcitol | Cholecalciferol | Placebo
Number analyzed (Participants) | 15 | 17 | 16
U/L | 87 (22) | 94 (24) | 101 (33)

3. Secondary Outcome: Serum Calcium
Description: This secondary outcome measure is change in serum calcium from baseline to final measure at 6 weeks differences in the 3 arms were compared
Time Frame: 6 weeks
Population: missing data from participant in paricalcitrol
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 15 | 17 | 16
mg/dL | 9.3 (0.3) | 9.4 (0.3) | 9.3 (0.6)

4. Secondary Outcome: Serum 25 OH Vitamin D
Description: This secondary outcome measure is change in serum hydroxy-vitaminD from baseline to final measure at 6 weeks differences in the 3 arms were compared
Time Frame: 6 weeks
Population: missing data from participant in paricalcitrol arm
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 15 | 17 | 16
ng/dL | 27 (7.2) | 38 (15) | 25 (7.8)

5. Secondary Outcome: Serum Phosphorus
Description: This secondary outcome measure is change in serum phosphorus from baseline to final measure at 6 weeks differences in the 3 arms were compared
Time Frame: 6 weeks
Population: missing data from all 3 participant arms
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 8 | 8 | 7
mg/dL | 4.0 (0.3) | 3.4 (0.5) | 3.7 (0.7)

6. Secondary Outcome: Osteocalcin
Description: This secondary outcome measure is change in osteocalcin from baseline to final measure at 6 weeks differences in the 3 arms were compared
Time Frame: 6 weeks
Population: Missing data from all 3 participant arms
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 14 | 15 | 16
ng/mL | 38 (21) | 39 (20) | 42 (21)

7. Secondary Outcome: N-Telopeptide Cross Linked Urine
Description: This secondary outcome measure is change in N-Telopeptide cross linked urine from baseline to final measure at 6 weeks, differences in the 3 arms were compared
Time Frame: 6 weeks
Population: Missing data from cholecalciferol and placebo participant arms
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 16 | 16 | 15
nmol | 74 (29) | 67 (34) | 77 (36)

8. Secondary Outcome: Bone Specific Alkaline Phosphatase
Description: This secondary outcome measure is change in bone specific alkaline phosphatase from baseline to final measure at 6 weeks, differences in the 3 arms were compared
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 15 | 15 | 16
u/L | 15 (4.8) | 19 (7.0) | 18 (5.0)

9. Secondary Outcome: 24 Hour Urine Calcium
Description: This secondary outcome measure is change in 24-hour urine calcium from baseline to final measure at 6 weeks, differences in the 3 arms were compared
Time Frame: 6 weeks
Population: Missing data from paricalcitol and cholecalciferol arms
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Paricalcitrol | Cholecalciferol | Placebo-controlled
Number analyzed (Participants) | 15 | 15 | 16
mg/dL | 132 (126) | 101 (111) | 135 (81)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Paricalcitriol: Paricalcitriol 1 mcg per day 7 days per week
- Cholecalciferol: cholecalciferol 5000 units per day, 7 days per week
- Placebo: Placebo capsules, one a day 7 days per week
Arm/Group | Paricalcitriol | Cholecalciferol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/16

LIMITATIONS AND CAVEATS:
The impact of malabsorption noted in Gastric Bypass patients may impact drug and nutritional absorption differently between patients and this effect can wane over time for some. Additionally, the study N and the short duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No